CLINICAL TRIAL: NCT05961345
Title: The Effect of Early Mobilization on Pain Level After Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cansel Bozer, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-01
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Mobilization; Pain; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity; Pain

STUDY DESIGN:
Intervention Model Description: two groups, a control and an experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: the experimental group was conducted early by the researcher and the outcome evaluations were performed by the researcher who blinded the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early mobilization (Experimental): The patients in the experimental group were mobilized at the 4th postoperative hour.
  Interventions: Other: late mobilization
- control group (late mobilization) (No Intervention): The patients in the control group were mobilized at the 6th hour as in the routine of the clinic.

INTERVENTIONS:
Other: late mobilization — Early mobilization of patients after surgery is supported. The relationship between early mobilization and pain level was examined. The experimental group is 80 people.
  Other Names: Early mobilization of patients after surgery is supported. The relationship between early mobilization and pain level was examined. The experimental group is 80 people.
  Arms: early mobilization

SUMMARY:
According to the definition of the WHO, obesity is the abnormal or excessive accumulation of fat in the body. Laparoscopic operations; It is a popular choice for bariatric surgery. A study is planned to determine postoperative early mobilization, postoperative pain and hospital stay in patients hospitalized in Bariatric Surgery post-operative clinics.

DETAILED DESCRIPTION:
According to the definition of the World Health Organization (WHO), obesity is the abnormal or excessive accumulation of fat in the body to the extent that it adversely affects health. Obesity; It is a chronic disease associated with multiple pathologies such as diabetes mellitus, cardiovascular diseases and different types of cancer, affecting the individual physically and psychosocially, which may occur due to social-economic level, lifestyle, cultural factors, and the decrease in energy consumption due to the slowing of the metabolic rate due to aging. Obesity is one of the serious and high prevalence health problems of the 21st century. When WHO data is examined; There are 1.9 billion overweight people and 650 million obese individuals in the world. When Turkey's data is analyzed, it ranks first in Europe with a 32 percent obesity rate.

Since obesity is preventable and treatable, many treatment protocols are available. In the treatment of obesity, it is planned to increase physical activities in addition to changing nutritional habits as the primary method. Subsequently, behavioral and medical treatment are among the preferred methods. If the desired result cannot be obtained, invasive or minimally invasive techniques are used in the treatment of this patient group with a body mass index (BMI) ≥ 40 kg/m2 or a BMI range of 35-39.9 kg/m2 and in addition to obesity-related metabolic diseases. bariatric surgery is considered.

Laparoscopic operations; It is a popular choice for bariatric surgery because of its ease of procedure, with proven long-term results in improving weight loss and obesity-related comorbidities. With the inclusion of the laparoscopic approach in surgical procedures, minimally invasive laparoscopic bariatric surgeries have become widespread in the field of bariatric surgery. Bariatric operations are associated with their unique short-term and long-term nutritional and procedural complications.

Enhanced Recovery After Surgery (ERAS), is patient recovery protocols (eras) that aim to minimize postoperative complications in patients and plan discharge in a short time. The basic principle of ERAS protocols; Reducing the pain associated with the stress and postoperative complications secondary to surgery, and ensuring the well-being of the patient by providing early mobilization in the postoperative period. After laparoscopic bariatric surgery, shoulder pain due to increased intra-abdominal pressure, stretching of the peritoneum, inability to take air given carbon dioxide (CO2), diaphragm irritation due to tension of muscle fibers, and visceral pain due to the interference of trocars on the abdominal wall after intra-abdominal intervention are observed.Unwillingness to mobilize and insufficient respiratory function can be seen in patients due to abdominal and shoulder pain.Muscle atrophy develops with the increase in insulin resistance in patients due to the prolonged postoperative immobilization time. In addition, the risk of thromboembolism should be considered.

It is planned to return the gastrointestinal functions of the patients after the surgery, to perform early muscle activities, to provide early venous conversion, to minimize the risks such as embolism, and early mobilization of the patients is supported. Although early mobilization causes these positive results, there is no study in the literature with the effectiveness of mobilization for postoperative pain. In addition, it is not known where the pain scales of the patients become stable in terms of postoperative discharge times. Therefore, our study has two main endpoints. It is planned that the study will guide the literature.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Can speak Turkish
* Agreeing to participate in the study
* No postoperative complications
* Patients with American Society of Anesthesiology (ASA) evaluation I, II, III were included in the sample group

Exclusion Criteria:

* Can not speak Turkish
* Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The Numerical Pain Rating Acale (NRS) | 72 hours
  Numerical pain rating scale is a scale that evaluates the severity of pain from 0 to 10.As the severity of pain increases, the number value increases. A number value of 0 means no pain, while 10 is the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Cansel Bozer, Principal Investigator — Cukurova University
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No